CLINICAL TRIAL: NCT03540615
Title: Randomized, Placebo-controlled, Double-blind Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Increasing Single Oral Doses of BAY1830839 in Healthy Male Subjects
Brief Title: BAY1830839: First in Man, Single Dose Escalation, Safety & Tolerability and Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 19150; 2017-001496-23 (EudraCT Number)
Record Dates: First submitted 2018-05-15; First posted 2018-05-30 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Dose escalation with safety assessment following each dose step.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAY1830839 (Experimental): Single Dose escalations
  Interventions: Drug: BAY1830839
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1830839 — Dose escalation in healthy male subjects
  Arms: BAY1830839
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to investigate

* the safety and tolerability of increasing single oral doses of BAY 1830839 versus placebo under fasted conditions
* the pharmacokinetics after single ascending oral doses of BAY 1830839 under fasted conditions

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) : ≥18.5 and ≤30 kg/m*2

Exclusion Criteria:

* Relevant diseases within the last 4 weeks prior to the first study drug administration
* Febrile illness within 4 weeks before the first study drug administration
* Known hypersensitivity to the study drugs or components of the preparations
* Clinically relevant findings in the physical examination

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
AUC of BAY1830839 in plasma | Day 1, 2, 3, 4, 6 ,7, 9, and 12
  AUC: area under the plasma concentration vs time curve from zero to infinity after single dose.
Cmax of BAY1830839 in plasma | Day 1, 2, 3, 4, 6 ,7, 9, and 12
  maximum observed drug concentration in plasma after single dose administration
Frequency of treatment-emergent adverse events | From first application of study intervention up to 30 days after end of treatment
Severity of treatment-emergent adverse events | From first application of study intervention up to 30 days after end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/